CLINICAL TRIAL: NCT00342628
Title: Evaluation of the Safety, Immunogenicity and Compatibility With DTP of an Investigational Vi-rEPA Conjugate Vaccine for Typhoid Fever When Administered to Infants in Vietnam Concurrently With DTP
Brief Title: Safety, Immunogenicity and Compatibility With DTP of a Typhoid Fever Vaccine in Infants
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 999999050; OH99-CH-N050 (Registry Identifier: NICHD IRB)
Record Dates: First submitted 2006-06-19; First posted 2006-06-21 (Estimated); Results first posted 2012-06-27 (Estimated); Last update posted 2012-06-27 (Estimated); Status verified 2012-05

CONDITIONS: Typhoid Fever
Keywords: Antibody; Reactions; Vaccine; Conjugate Vaccine; Typhoid Fever; Trial; Safety; Immunogenicity; Comparability; DTP
MeSH Terms: conditions — Typhoid Fever | interventions — Haemophilus influenza type b polysaccharide vaccine-tetanus toxin conjugate

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Vi-rEPA plus DTP (Experimental): Vi-rEPA and DTP at 2, 4, 6 months, and Vi-rEPA at 12 months
  Interventions: Biological: Vi-rEPA conjugate vaccine for typhoid fever; Biological: DTP
- Hib-TT plus DTP (Active Comparator): Hib-TT and DTP at 2,4 and 6 months, Hib-TT at 12 months
  Interventions: Biological: Hib-TT; Biological: DTP
- EPI (Active Comparator): DTP at 2,4 and 6 months
  Interventions: Biological: DTP

INTERVENTIONS:
Biological: Vi-rEPA conjugate vaccine for typhoid fever — Vi-rEPA contains a 25 ug/dose of Vi (Sanofi-Pasteur Lot 130) and rEPA in 0.2 N NaCl, 10 mM phosphate PH 7.2 and 0.01% thimerosal.
  Other Names: Vi conjugate
  Arms: Vi-rEPA plus DTP
Biological: Hib-TT — Hib-TT is Hemophilus influenzae type b-tetanus toxoid conjugate vaccine (ActHib, NDC#49281-545-05 Sanofi-Pasteur, France) in single-dose vials containing 10 ugof Hib CP conjugated to 24 ug of tetanus toxoid
  Other Names: Hib conjugate
  Arms: Hib-TT plus DTP
Biological: DTP — DTP, diphtheria, tetanus toxoid and pertussis vaccine were from the Ministry of Health, Vietnam for routine infant immunization
  Other Names: EPI vaccine

SUMMARY:
The purpose of this study is to evaluate the safety, immunogenicity, and compatibility of our Vi-rEPA conjugate administered to infants with their routine vaccinations.

We propose to recruit 300 full term healthy newborns in Vietnam and randomly divide them to receive Vi-rEPA plus DTP, Hib-TT (not yet used in Vietnam) plus DTP, or DTP alone. Consent is obtained following interviews of mothers during prenatal visits, or after delivery. All vaccines will be administered at 2, 4, and 6 months. A booster of Vi-rEPA or Hib-TT conjugate will be administered at 12 months of age and reactions monitored at 6, 24 and 48 hours after each injection. Maternal and cord blood samples are collected during labor and at delivery. Blood will be taken at 7, and 12 months of age from all study infants and at 13 months from infants injected with Vi-rEPA or with Hib-TT at 12 months. The blood samples will be assayed for Vi, Hib, diphtheria, tetanus and pertussis antibodies.

The levels of serum IgG anti-Vi elicited by Vi-rEPA administered to infants by the above schedule will be compared to those elicited by this vaccine in 2 to 5 year-olds in the efficacy trial conducted in Dong Thap Province, Vietnam.

DETAILED DESCRIPTION:
Typhoid fever remains common, serious, and difficult-to-treat throughout the world including Vietnam. Limitations of the three licensed typhoid vaccines have prevented their use for routine vaccination of infants. The most recent, Vi polysaccharide typhoid vaccine is useful only in individuals greater than or equal to 5 years of age because of its age-related and T-cell independent properties. The immunogenicity of Vi in individuals less than 5 years-old has been improved by binding it to a protein. In 2 to 4-year-olds, 2 injections of the Vi conjugate induced higher levels of serum IgG anti-Vi than Vi in 5 to 14-year-olds.

A double-blind, placebo controlled and randomized efficacy study in 2 -to-5 years old children in Vietnam showed an over-all efficacy after 27 months of active surveillance followed by 19 months of passive surveillance of 89%. Subsequently a dosage study in the same age group showed the highest antibody levels were induced by the 25 mcg dose.

Now we wish to evaluate the safety, immunogenicity, and compatibility of our Vi-rEPA conjugate administered to infants with their routine vaccinations.

We propose to recruit 300 full term healthy newborns in Vietnam and randomly divide them to receive Vi-rEPA plus DTP (Group A), Hib-TT (not yet used in Vietnam) plus DTP (Group B), or DTP alone (Group C). Maternal and cord blood are taken routinely on all deliveries in Vietnam; these sera will be retrieved for storage when consent is obtained following interviews of mothers during prenatal visits, or after delivery. All vaccines will be administered at 2, 4, and 6 months. A booster of Vi-rEPA or Hib-TT conjugate will be administered at 12 months of age and reactions monitored at 6, 24 and 48 hours after each injection. Blood will be taken at 7, and 12 months of age from all study infants and at 13 months from infants injected with Vi-rEPA or with Hib-TT at 12 months. The blood samples will be assayed for Vi, Hib, diphtheria, tetanus and pertussis antibodies.

The levels of serum IgG anti-Vi elicited by Vi-rEPA administered to infants by the above schedule will be compared to those elicited by this vaccine in 2 to 5 year-olds in the efficacy trial conducted in Dong Thap.

ELIGIBILITY:
Inclusion criteria:

* Healthy full-term newborns.
* Birth weights of >=2500 grams.

Exclusion criteria:

* Newborns without maternal and cord blood samples
* Newborns born to mothers with serious medical problems.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 301 (Actual)
Dates: Start 2006-07; Primary Completion 2008-04 (Actual); Study Completion 2011-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Feng-Ying (Kimi) Lin, MD, MPH, Study Director — PDMI, NICHD, NIH
Locations (1):
- Thanh Thuy District Health Center, Việt Trì, Phu Tho, Vietnam

REFERENCES:
- [Background] Acharya IL, Lowe CU, Thapa R, Gurubacharya VL, Shrestha MB, Cadoz M, Schulz D, Armand J, Bryla DA, Trollfors B, et al. Prevention of typhoid fever in Nepal with the Vi capsular polysaccharide of Salmonella typhi. A preliminary report. N Engl J Med. 1987 Oct 29;317(18):1101-4. doi: 10.1056/NEJM198710293171801. PMID 3657877
- [Background] Crump JA, Mintz ED. Global trends in typhoid and paratyphoid Fever. Clin Infect Dis. 2010 Jan 15;50(2):241-6. doi: 10.1086/649541. PMID 20014951
- [Background] Gilman RH, Terminel M, Levine MM, Hernandez-Mendoza P, Hornick RB. Relative efficacy of blood, urine, rectal swab, bone-marrow, and rose-spot cultures for recovery of Salmonella typhi in typhoid fever. Lancet. 1975 May 31;1(7918):1211-3. doi: 10.1016/s0140-6736(75)92194-7. PMID 48834
- [Background] Klugman KP, Gilbertson IT, Koornhof HJ, Robbins JB, Schneerson R, Schulz D, Cadoz M, Armand J. Protective activity of Vi capsular polysaccharide vaccine against typhoid fever. Lancet. 1987 Nov 21;2(8569):1165-9. doi: 10.1016/s0140-6736(87)91316-x. PMID 2890805
- [Background] Kossaczka Z, Lin FY, Ho VA, Thuy NT, Van Bay P, Thanh TC, Khiem HB, Trach DD, Karpas A, Hunt S, Bryla DA, Schneerson R, Robbins JB, Szu SC. Safety and immunogenicity of Vi conjugate vaccines for typhoid fever in adults, teenagers, and 2- to 4-year-old children in Vietnam. Infect Immun. 1999 Nov;67(11):5806-10. doi: 10.1128/IAI.67.11.5806-5810.1999. PMID 10531232
- [Background] Mai NL, Phan VB, Vo AH, Tran CT, Lin FY, Bryla DA, Chu C, Schiloach J, Robbins JB, Schneerson R, Szu SC. Persistent efficacy of Vi conjugate vaccine against typhoid fever in young children. N Engl J Med. 2003 Oct 2;349(14):1390-1. doi: 10.1056/NEJM200310023491423. No abstract available. PMID 14523155
- [Background] Levine MM, Ferreccio C, Abrego P, Martin OS, Ortiz E, Cryz S. Duration of efficacy of Ty21a, attenuated Salmonella typhi live oral vaccine. Vaccine. 1999 Oct 1;17 Suppl 2:S22-7. doi: 10.1016/s0264-410x(99)00231-5. PMID 10506405
- [Background] Lin FY, Vo AH, Phan VB, Nguyen TT, Bryla D, Tran CT, Ha BK, Dang DT, Robbins JB. The epidemiology of typhoid fever in the Dong Thap Province, Mekong Delta region of Vietnam. Am J Trop Med Hyg. 2000 May;62(5):644-8. doi: 10.4269/ajtmh.2000.62.644. PMID 11289678
- [Background] Lin FY, Ho VA, Khiem HB, Trach DD, Bay PV, Thanh TC, Kossaczka Z, Bryla DA, Shiloach J, Robbins JB, Schneerson R, Szu SC. The efficacy of a Salmonella typhi Vi conjugate vaccine in two-to-five-year-old children. N Engl J Med. 2001 Apr 26;344(17):1263-9. doi: 10.1056/NEJM200104263441701. PMID 11320385
- [Background] Ochiai RL, Acosta CJ, Danovaro-Holliday MC, Baiqing D, Bhattacharya SK, Agtini MD, Bhutta ZA, Canh DG, Ali M, Shin S, Wain J, Page AL, Albert MJ, Farrar J, Abu-Elyazeed R, Pang T, Galindo CM, von Seidlein L, Clemens JD; Domi Typhoid Study Group. A study of typhoid fever in five Asian countries: disease burden and implications for controls. Bull World Health Organ. 2008 Apr;86(4):260-8. doi: 10.2471/blt.06.039818. PMID 18438514
- [Background] Sinha A, Sazawal S, Kumar R, Sood S, Reddaiah VP, Singh B, Rao M, Naficy A, Clemens JD, Bhan MK. Typhoid fever in children aged less than 5 years. Lancet. 1999 Aug 28;354(9180):734-7. doi: 10.1016/S0140-6736(98)09001-1. PMID 10475185
- [Background] Szu SC, Stone AL, Robbins JD, Schneerson R, Robbins JB. Vi capsular polysaccharide-protein conjugates for prevention of typhoid fever. Preparation, characterization, and immunogenicity in laboratory animals. J Exp Med. 1987 Nov 1;166(5):1510-24. doi: 10.1084/jem.166.5.1510. PMID 3681191
- [Background] Taylor DN, Levine MM, Kuppens L, Ivanoff B. Why are typhoid vaccines not recommended for epidemic typhoid fever? J Infect Dis. 1999 Dec;180(6):2089-90. doi: 10.1086/315159. No abstract available. PMID 10558978

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Informed consent was obtained from expectant women during prenatal visits in Thanh Thuy District, Phu-Tho Province, Vietnam. Mothers and newborns were enrolled during labor at commune/district health centers from July 26, 2006 to March 8, 2007. Only fullterm newborns with birth weights of >=2500 grams were enrolled.
Groups:
- Vi-rEPA Plus DTP: Vi-rEPA plus DTP at 2, 4, 6 and Vi-rEPA at 12 months of age
- Hib-TT Plus DTP: Hib-TT plus DTP at 2,4,6 and Hib-TT at 12 months of age
- DTP Vaccines: DTP at 2, 4, and 6 months of age
Period: Overall Study
Arm/Group | Vi-rEPA Plus DTP | Hib-TT Plus DTP | DTP Vaccines
Started | 100 | 101 | 100
Completed | 80 (84 completed 4 injections, 4 were lost-to-followup after the 4th injection) | 80 (83 completed 4 injections, 3 were lost-to-followup after 4th injection) | 81 (97 completed 3 injections of DTP alone, 16 were lost-to-followup for blood drawing at 12 months.)
Not Completed | 20 | 21 | 19
Not completed — Withdrawal by Subject | 19 | 19 | 18
Not completed — Death | 1 | 1 | 0
Not completed — moved residence | 0 | 1 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Vi-rEPA Plus DTP | Hib-TT Plus DTP | DTP Vaccines | Total
Number analyzed (Participants) | 100 | 101 | 100 | 301
Age, Customized [Mean (Full Range); unit: Days] — Study participants are infants recruited at birth, injected with experimental and comparison vaccine at 2, 4, 6 and 12 months of age.
  Days
    Age at 1st injection | 77 [61 to 92] | 76 [61 to 92] | 76 [61 to 92] | 77 [61 to 92]
    Age at 2nd injection | 137 [121 to 151] | 137 [120 to 154] | 137 [121 to 151] | 137 [120 to 154]
    Age at 3rd injection | 197 [181 to 212] | 198 [182 to 211] | 197 [181 to 211] | 197 [181 to 212]
    Age at 4th injection | 382 [365 to 420] | 381 [365 to 406] | NA [NA to NA] — No injection given | 382 [365 to 420]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 52 | 53 | 46 | 151
  Male | 48 | 48 | 54 | 150

OUTCOME MEASURES:

1. Primary Outcome: Number of Infants With Adverse Reactions After Vaccination
Description: Number of infants with Fever>=38.0 C, Induration>=2.5cm at DTP site, Induration>=2.5cm,Vi-rEPA/Hib-TT site, Erythema>=2.5cm, at DTP site, Erythema>=2.5cm, Vi-rEPA/Hib-TT site, Inconsolable crying<4hr, Inconsolable crying>=4hr per injection with Vi conjugate vaccine given in conjunction with DTP in infants.
Time Frame: at 2, 4, 6 and 12 months
Population: The number of infants injected in each group for each injection was used to determine the rate of adverse reactions.
Measure: Number; unit: participants
Arm/Group | Vi-rEPA Plus DTP | Hib-TT Plus DTP | DTP Vaccines
Number analyzed (Participants) | 100 | 101 | 100
participants
  Fever>=38.0 C 1st inj | 22 | 24 | 17
  Fever>=38.0 C 2nd inj | 7 | 7 | 6
  Fever>=38.0 C 3rd inj | 4 | 2 | 0
  Fever>=38.0 C 4th inj | 2 | 0 | NA — no injection for this group
  Induration>=2.5cm, at DTP site, Inj 1 | 2 | 2 | 5
  Induration>=2.5cm, at DTP site, Inj 2 | 1 | 1 | 2
  Induration>=2.5cm, at DTP site, Inj 3 | 0 | 0 | 0
  Induration>=2.5cm, at DTP site, Inj 4 | NA — No injection for this group | NA — no injection for this group | NA — no injection for this group
  Induration>=2.5cm,Vi-rEPA/Hib-TT site, Inj 1 | 1 | 0 | NA — no Vi-rEPA/Hib-TT site for this group
  Induration>=2.5cm,Vi-rEPA/Hib-TT site, Inj 2 | 0 | 0 | NA — no Vi-rEPA/Hib-TT site for this group
  Induration>=2.5cm,Vi-rEPA/Hib-TT site, Inj 3 | 0 | 0 | NA — no Vi-rEPA/Hib-TT site for this group
  Induration>=2.5cm,Vi-rEPA/Hib-TT site, Inj 4 | 0 | 0 | NA — no Vi-rEPA/Hib-TT site for this group
  Erythema>=2.5cm, at DTP site, Inj 1 | 3 | 1 | 4
  Erythema>=2.5cm, at DTP site, Inj 2 | 0 | 0 | 0
  Erythema>=2.5cm, at DTP site, Inj 3 | 0 | 0 | 0
  Erythema>=2.5cm, at DTP site, Inj 4 | NA — No injection for this group | NA — no injection for this group | NA — no injection for this group
  Erythema>=2.5cm, Vi-rEPA/Hib-TT site, Inj 1 | 2 | 0 | NA — no Vi-rEPA/Hib-TT site for this group
  Erythema>=2.5cm, Vi-rEPA/Hib-TT site, Inj 2 | 0 | 0 | NA — no Vi-rEPA/Hib-TT site for this group
  Erythema>=2.5cm, Vi-rEPA/Hib-TT site, Inj 3 | 0 | 0 | NA — no Vi-rEPA/Hib-TT site for this group
  Erythema>=2.5cm, Vi-rEPA/Hib-TT site, Inj 4 | 0 | 0 | NA — no Vi-rEPA/Hib-TT site for this group
  Inconsolable crying<4hr, inj 1 | 5 | 7 | 2
  Inconsolable crying<4hr, inj 2 | 0 | 0 | 0
  Inconsolable crying<4hr, inj 3 | 0 | 0 | 0
  Inconsolable crying<4hr, inj 4 | 0 | 0 | NA — no injection for this group
  Inconsolable crying>=4hr, inj 1 | 2 | 1 | 0
  Inconsolable crying>=4hr, inj 2 | 0 | 0 | 0
  Inconsolable crying>=4hr, inj 3 | 0 | 0 | 0
  Inconsolable crying>=4hr, inj 4 | 0 | 0 | NA — no injection for this group

2. Secondary Outcome: IgG Anti-Vi Levels
Description: IgG anti-Vi was measured by ELISA and expressed as ELISA units (EU)in all sera.
Time Frame: cord sera, infants' sera at 7, 12 and 13 months
Population: Only participants with available cord sera are included in the analyses
Measure: Geometric Mean (Inter-Quartile Range); unit: ELISA units
Arm/Group | Vi-rEPA Plus DTP | Hib-TT Plus DTP | DTP Vaccines
Number analyzed (Participants) | 100 | 100 | 100
ELISA units
  IgG anti-Vi (cord sera) | 0.66 [0.30 to 1.46] | 0.55 [0.26 to 1.02] | 0.52 [0.20 to 0.98]
  IgG anti-Vi at 7 months | 17.42 [7.33 to 47.25] | 0.16 [0.10 to 0.25] | 0.05 [0.02 to 0.09]
  IgG anti-Vi at 12 months | 4.76 [2.20 to 12.71] | 0.17 [0.11 to 0.27] | 0.04 [0.02 to 0.08]
  IgG anti-Vi at 13 months | 50.07 [22.33 to 133.61] | 0.19 [0.11 to 0.27] | NA [NA to NA] — No serum samples were collected for this group

3. Secondary Outcome: Antibody Responses to Tetanus Toxoid, Diphtheria Toxoid, and Pertussis Toxin
Description: IgG anti-diphtheria toxoid (DT), -tetanus toxoid (TT) and -pertussis toxin (PT) were measured by ELISA in sera of 30 randomly chosen infants per group.
Time Frame: Cord sera, and infants' sera at 7, 12 and 13 months of age
Population: Randomly chosen 30 participants in each group. Four in Comparison group 2 were excluded from analyses due to classification error.
Measure: Geometric Mean (Inter-Quartile Range); unit: U/ml
Arm/Group | Vi-rEPA Plus DTP | Hib-TT Plus DTP | DTP Vaccines
Number analyzed (Participants) | 30 | 30 | 26
U/ml
  Anti-TT (U/ml) cord sera | 4.81 [2.94 to 10.62] | 3.92 [1.98 to 7.58] | 4.37 [1.01 to 12.91]
  Anti-TT (U/ml) at 7 months | 4.18 [3.18 to 6.97] | 5.16 [3.16 to 8.32] | 4.03 [2.78 to 5.28]
  Anti-TT (U/ml) at 12 months | 0.46 [0.36 to 0.69] | 0.87 [0.73 to 1.17] | 0.53 [0.37 to 0.74]
  Anti-TT (U/ml) at 13 months | 0.39 [0.31 to 0.56] | 5.15 [2.85 to 12.01] | NA [NA to NA] — No blood samples collected at 13 months
  Anti-DT (U/ml) cord sera | 8.29 [6.20 to 14.13] | 8.63 [4.39 to 16.65] | 11.84 [6.14 to 15.94]
  Anti-DT (U/ml) at 7 months | 62.10 [42.25 to 96.58] | 74.56 [34.93 to 152.93] | 55.79 [41.18 to 97.30]
  Anti-DT (U/ml) at 12 months | 8.27 [5.62 to 13.24] | 10.07 [4.95 to 18.78] | 9.10 [5.60 to 15.68]
  Anti-DT (U/ml) at 13 months | 7.93 [6.06 to 11.19] | 8.66 [4.33 to 15.42] | NA [NA to NA] — No blood samples collected at 13 months.
  Anti-PT (U/ml) cord sera | 26.58 [18.04 to 38.86] | 33.71 [22.62 to 54.55] | 25.30 [18.36 to 39.67]
  Anti-PT (U/ml) at 7 months | 199.72 [125.36 to 522.88] | 311.91 [166.06 to 467.77] | 283.67 [156.11 to 554.64]
  Anti-PT (U/ml) at 12 months | 30.86 [20.38 to 77.06] | 41.03 [19.86 to 73.04] | 42.94 [28.31 to 71.89]
  Anti-PT (U/ml) at 13 months | 25.86 [14.89 to 51.21] | 33.52 [14.51 to 70.22] | NA [NA to NA] — No blood samples collected at 13 months

4. Secondary Outcome: Antibody Responses to Hib CP
Description: IgG anti-Hib CP was measured by ELISA in sera of 30 randomly chosen infants per group
Time Frame: Cord sera and infant sera at 7, 12, and 13 months
Population: as for outcome 3
Measure: Geometric Mean (Inter-Quartile Range); unit: mcg/ml
Arm/Group | Vi-rEPA Plus DTP | Hib-TT Plus DTP | DTP Vaccines
Number analyzed (Participants) | 30 | 30 | 30
mcg/ml
  Anti-Hib CP (mcg/ml) cord sera | 2.11 [0.99 to 3.95] | 1.33 [0.75 to 3.18] | 2.0 [0.87 to 3.90]
  Anti-Hib CP (mcg/ml) at 7 months | 0.32 [0.11 to 0.53] | 8.35 [2.95 to 29.65] | 0.33 [0.20 to 0.38]
  Anti-Hib CP (mcg/ml) at 12 months | 0.29 [0.09 to 1.23] | 1.79 [0.98 to 3.21] | 0.37 [0.20 to 0.52]
  Anti-Hib CP (mcg/ml) at 13 months | 0.29 [0.09 to 1.04] | 24.53 [10.23 to 68.26] | NA [NA to NA] — No blood samples were collected at 13 months

ADVERSE EVENTS:
Time Frame: 2, 4, 6 and 12 months
Description: Vaccinees were visited by health care workers at 6 hours, one and two days after each injection for measurements of temperature, inspection of injection site and record other systemic reactions.
Arm/Group | Vi-rEPA Plus DTP | Hib-TT Plus DTP | DTP Vaccines
Serious Adverse Events (participants affected / at risk) | 1/100 | 1/101 | 0/100
Other Adverse Events (participants affected / at risk) | 0/100 | 0/101 | 0/100
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Vi-rEPA Plus DTP (N=100) | Hib-TT Plus DTP (N=101) | DTP Vaccines (N=100)
Death (General disorders) | 1 (1) | 1 (1) | 0 (0) — A 5 month old injected 1 X with Vi-rEPA died of septicemia post surgery for "nonfunctioning" kidneys. A 4 month old died of pneumonia after 2nd injection of Hib-TT. Deaths were unrelated to study, noted only because they affect the participant flow.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes